CLINICAL TRIAL: NCT01805765
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Clinical Trial on the Effects of Chinese Medicine Formula (Qing'E) on Menopausal Symptoms
Brief Title: Qing'E Formula Therapy on Menopausal Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Longhua Hospital (Other); Shanghai Yueyang Integrated Medicine Hospital (Other); Shanghai Municipal Hospital of Traditional Chinese Medicine (Other); Shanghai Putuo District Center Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QE-2458-1; SHU-5366432 (Other: Shanghai University of TCM)
Record Dates: First submitted 2013-02-26; First posted 2013-03-06 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2013-03

CONDITIONS: Menopause
Keywords: menopausal syndrome; climacteric syndrome; Hot flashes; Sweat
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qing'E pills (Active Comparator): 9 g pills,twice a day for 12 weeks
  Interventions: Drug: Qing'E pills
- Placebo (Placebo Comparator): 9 g pills,twice a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Qing'E pills — composed of eucommia, psoralen, walnuts and garlic
  Arms: Qing'E pills
Drug: Placebo — Containing 2% of Qing'E pills
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate whether a Chinese medicine formula (Qing'E) is effective in alleviating menopausal symptoms and safety.

DETAILED DESCRIPTION:
This is a double-blind placebo-controlled randomized clinical trial to evaluate whether a Chinese medicine formula (Qing'E, composed of eucommia, psoralen, walnuts and garlic) is effective in alleviating menopausal symptoms. 240 Chinese women with menopausal symptoms will be recruited and randomized into two groups. One is treatment group with 12 weeks of Qing'E pills (well-controlled), the other is controlled group with 12 weeks of placebo. The treatment outcome measures include: 1) the severity of menopausal symptoms: self-recording of daily frequency of vasomotor symptoms (hot flushes), the Kupperman index. 2) NEI network indices. 3) Urine metabolomics. All measures are conducted at baseline and endpoint except the self-recoding of vasomotor symptoms, Kupperman index and urine metabolomics. Tyhe investigators expect this research will provide an effective and safe therapy for menopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Women age between 40 to 60 Years, Suffering from irregular menstrual cycle or amenorrhea of 3-11 months.
2. Moderate to severe hot flashes (associated with sweating)≥5 times /24 hours.
3. Patients unused estrogen tablets or progesterone injection in 6 months.
4. Patients must discontinue other therapies in the treatment of menopausal syndrome for more than 3 months.
5. Get subjects informed consent process should comply with GCP requirements.

Exclusion Criteria:

1. Patients with hypertension, primary hypotension and chronic anemia (Hb ≤ 90 g / L).
2. Bilateral oophorectomy, endometrial lesions, uterine polyps, abnormal vaginal bleeding, severe breast hyperplasia, with family history of breast cancer.
3. Allergic constitution and known allergy to the drug.
4. Patients with diseases of the cardiovascular, cerebrovascular, liver, kidney and hematopoietic system, or mentally ill.
5. Patients with hyperthyroidism, coronary atheroma, diabetes, obesity (body mass index of more than 30 kg/m2), migraine, malignant tumors, thromboembolic disease, gastrointestinal diseases affect absorption or autoimmune diseases.
6. Alcoholics or smokers (past or smoking).
7. Patients are participating in other clinical trials.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hot flushes | 12 weeks
  Change in frequency of hot flushes from baseline to week 12.

SECONDARY OUTCOMES:
Hot flushes | 4 weeks, 8 weeks
  Change in frequency of hot flushes from baseline to week 4 and week 8.
Hot flushes | 4 weeks, 8 weeks and 12 weeks
  Decline rate of hot flushes from baseline to week 4, week 8 and week 12;
Mean differences of Kupperman index | 4 weeks, 8 weeks and 12 weeks
  To calculate the Kupperman index, the symptoms were weighted as follows: hot flashes (4), insomnia (2), nervousness (2), and all other symptoms (night sweats, depressed mood (melancholy), dizziness, tiredness, joint and muscular pain, headache, and palpitations (1). The highest potential score is thus 51. The score of hot flashes was based on number of complaints per day: slight (more than 5), moderate (5-10), and severe (more than 10)
Mean difference of single clinical symptom in Kupperman index | 12 weeks

OTHER OUTCOMES:
Nerve-endocrine-immune (NEI） network profile | 12 weeks
  To evaluate the difference of NEI network expression from baseline to 12 weeks. The indices in NEI network include:
  Hypothalamic-pituitary-adrenal axis: CRH, ATCH, CORT; Hypothalamic-pituitary-thyroid axis: TRH, T3, T4; Renin - angiotensin - aldosterone system: PRA, Ang2, ALD; Sex hormones: E2, FSH; Immune factors: TNF-α、IL-6、IL-1; Cardiovascular indicators: ET, NO, Hcy, Folic acid
Urine metabolomics | 4 weeks, 8 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qingshan Zheng, Doctor, Study Chair — Shanghai Universitu of TCM
Locations (1):
- Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China